CLINICAL TRIAL: NCT02161653
Title: Impact of Metadoxine in the Oxidative Stress and Early Mortality in Patients With Severe Alcoholic Hepatitis
Brief Title: Metadoxine as a Therapy for Severe Alcoholic Hepatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital General de Mexico (Other Government)
Responsible Party: Principal Investigator, MARIA DE FATIMA HIGUERA DE LA TIJERA, MD, MSc., Hospital General de Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DI/10/107/3/43
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2014-11-11 (Estimated); Status verified 2014-11

CONDITIONS: Severe Alcoholic Hepatitis
Keywords: Severe alcoholic hepatitis; survival; oxidative stress
MeSH Terms: conditions — Hepatitis, Alcoholic | interventions — Prednisone; metadoxine; Pentoxifylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Prednisone (No Intervention): Prednisone 40 mg daily by mouth during 30 days.
- Pentoxifylline (No Intervention): Pentoxifylline 400 mg thrice in day by mouth during 30 days
- Prednisone plus metadoxine (Experimental): Prednisone 40 mg daily by mouth plus Metadoxine 500 mg thrice in day by mouth during 30 days.
  Interventions: Drug: Prednisone plus Metadoxine
- Pentoxifylline plus metadoxine (Experimental): Pentoxifylline 400 mg thrice in day by mouth plus Metadoxine 500 mg thrice in day by mouth during 30 days.
  Interventions: Drug: Pentoxifylline plus Metadoxine

INTERVENTIONS:
Drug: Prednisone plus Metadoxine
  Arms: Prednisone plus metadoxine
Drug: Pentoxifylline plus Metadoxine
  Arms: Pentoxifylline plus metadoxine

SUMMARY:
The purpose of this study is to determine whether metadoxine is effective for improve survival and reduced oxidative stress in patients with severe alcoholic hepatitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical and biochemical criteria for severe alcoholic hepatitis: Total bilirubin greater than 5 mg/dl in absence of biliary tract obstruction evidenced by ultrasound, history of chronic alcohol intake, leukocytosis, neutrophilia, elevation of transaminases with an aspartate aminotransferase / alanine aminotransferase ratio equal or greater than 2, discriminant function greater than 32.

Exclusion Criteria:

* Diabetes, chronic kidney disease, hepatitis C, hepatitis B and or human immunodeficiency virus infection, asthma or history of atopy or allergic reactions, therapy in the previous two years with steroids, pentoxifylline, metadoxine, S-adenosyl L- methionine, antioxidants or multivitamins.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2010-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
30 day-survival | 30 days
Malondialdehyde serum levels | 14 and 30 days

SECONDARY OUTCOMES:
3 month-survival | 3 months
6 month-survival | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General de Mexico, Mexico City, D.f., Mexico

REFERENCES:
- [Derived] Higuera-de la Tijera F, Servin-Caamano AI, Serralde-Zuniga AE, Cruz-Herrera J, Perez-Torres E, Abdo-Francis JM, Salas-Gordillo F, Perez-Hernandez JL. Metadoxine improves the three- and six-month survival rates in patients with severe alcoholic hepatitis. World J Gastroenterol. 2015 Apr 28;21(16):4975-85. doi: 10.3748/wjg.v21.i16.4975. PMID 25945012